CLINICAL TRIAL: NCT01704053
Title: Monitoring The Anticoagulatory Effects of Dabigatran and Rivaroxaban On Plasmatic and Cellular Coagulation by Rotational Thrombelastometry/-Graphy and Multiple Platelet Function Analyzer
Brief Title: Effect of New Oral Anticoagulants Dabigatran and Rivaroxaban on Point of Care Coagulation Testing - an Ex-Vivo Study
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Matthias Klages, M.D., Johann Wolfgang Goethe University Hospital
Other Study IDs: NOAPOC-271/12
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Clot Formation and Platelet Aggregation in Point of Care Testing
Keywords: New Oral Anticoagulants; Dabigatran; Rivaroxaban; Thrombelastometry/-graphy (ROTEM, TEG); Multiple Platelet Function Analyzer (Multiplate)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is determine whether point of care coagulation testing is able to map the anticoagulatory effects of new oral anticoagulants dabigatran and rivaroxaban. Used as devices are thrombelastometry/-graphy (ROTEM, TEG)and multiple platelet function analyzer (Multiplate).

DETAILED DESCRIPTION:
Patients receiving dabigatran or rivaroxaban in therapeutic doses are recruited. Blood will be taken twice in correlation to the time of drug intake (before and 3 hours after drug intake). The results of thrombelastometry/-graphy and multiple platelet function analyzer will be compared directly with the concentrations determined by plasma concentration assays.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Dabigatran or Rivaroxaban
* Adults > 18 years

Exclusion Criteria:

* Patients receiving concomittantly inhibitors of platelet function
* Renal insufficiency (Creatinine > 1,5 mg/dl), Urea > 80 mg/dl)
* Hemodialysis
* Hepatic Dysfunction (AST > 30 U/l, ALT > 30 U/l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic. Patients with non-valvular atrial fibrillation who receive Dabigatran or Rivaroxaban for prevention of stroke and systemic embolism.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of University hospital of Frankfurt/Main, Department of Anesthesiology, Intensive-Care Medicine and Pain Therapy, Frankfurt am Main, Hesse, Germany